CLINICAL TRIAL: NCT05328037
Title: Study on the Association Between Vitamin C Deficiency and Diarrhea in Children
Acronym: VITAL
Status: Completed | Type: Observational
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut Cochin (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-063; ID-RCB number : 2021-A00632-39 (Other: French national registration number of the study)
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Diarrhea; Infantile
Keywords: Vitamin C; Diarrhea; Children
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute diarrhea cases: Children with acute diarrhea defined as at least 3 loose or watery stools per day for at least 3 consecutive days and up to 10 consecutive days
  Interventions: Diagnostic Test: Blood sample collection
- Chronic diarrhea cases: Children with chronic diarrhea defined as 3 or more loose or liquid stools per day for at least 4 weeks
  Interventions: Diagnostic Test: Blood sample collection
- Controls: Children without fever or signs of infection or ongoing diarrhea
  Interventions: Diagnostic Test: Blood sample collection

INTERVENTIONS:
Diagnostic Test: Blood sample collection — Blood sample collection for dosage of vitamin C

SUMMARY:
Diarrheal disease is the second leading cause of death in children under five, althought it is both preventable and treatable. The causative factors of diarrheal diseases vary a lot from region to region (bacteria, viruses, parasites). Diarrhea is one of the main causes of malnutrition in children under five years of age. Inversely, nutritional deficiency, particularly vitamin C deficiency, can be a risk factor for diarrhea.

The main objective of this study is to assess the impact of vitamin C deficiency on diarrheal infection in children aged 2 to 5 years in countries with a high diarrheal rate. This pilot case-control study will be conducted in metropolitan France, Africa and South America. This question will be addressed by comparing vitamin C levels in children with diarrhea, regardless of the infectious agent, to levels in age- and sex-matched controls.

DETAILED DESCRIPTION:
Diarrheal disease is the second leading cause of death in children under five, althought it is both preventable and treatable. The causative factors of diarrheal diseases vary a lot from region to region (bacteria, viruses, parasites). Diarrhea is one of the main causes of malnutrition in children under five years of age. Inversely, nutritional deficiency, particularly vitamin C deficiency, can be a risk factor for diarrhea.

The main objective of this study is to assess the impact of vitamin C deficiency on diarrheal infection in children aged 2 to 5 years in countries with a high diarrheal rate. This pilot case-control study will be conducted in metropolitan France, Africa and South America. This question will be addressed by comparing vitamin C levels in children with diarrhea, regardless of the infectious agent, to levels in age- and sex-matched controls.

The study aims at (i) determining whether vitamin-deficiency may occurs in children living in developing countries and at (ii) determining the plasma vitamin A, C and E concentrations in children suffering of diarrheal diseases.

A total of 360 children will participate to the study.

ELIGIBILITY:
Controls :

Inclusion Criteria:

* not suffering of diarrhea
* no fever
* no sign of infection

Exclusion criteria :

* Suspected or diagnosed infectious diseases
* Known genetic diseases
* Known diseases that may interfere with iron and/or vitamin C metabolism
* Known inflammatory diseases
* Malnutrition
* Diarrhea
* Fever
* Positive malaria rapid diagnostic test (Africa)
* Child currently being breastfed

Chronic diarrhea cases :

Inclusion Criteria:

-Children suffering from chronic diarrhea defined by the emission of at least 3 soft or liquid stools per day for at least 4 weeks.

Exclusion criteria :

* Suspected or diagnosed infectious diseases
* Known genetic diseases
* Known diseases that may interfere with iron and/or vitamin C metabolism
* Known inflammatory diseases
* Positive malaria rapid diagnostic test (Africa)
* Antibiotic treatment prescribed within 10 days prior to sampling
* Nutritional supplements in the three months prior to sampling
* Vitamin C supplementation in the last 3 months prior to blood collection
* Child currently being breastfed

Acute diarrhea cases :

Inclusion Criteria:

-Children suffering from acute diarrhea defined as 3 or more loose or watery stools per day for at least 3 consecutive days and up to 10 consecutive days.

Exclusion criteria :

* Malnutrition
* Suspected or diagnosed infectious diseases
* Known genetic diseases
* Known diseases that may interfere with iron and/or vitamin C metabolism
* Known inflammatory diseases
* Positive malaria rapid diagnostic test (Africa)
* Antibiotic treatment prescribed within 10 days prior to sampling
* Nutritional supplements in the three months prior to sampling
* Vitamin C supplementation in the last 3 months prior to blood collection
* Child currently being breastfed

Ages: 18 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population is children aged 18 months to 5 years (60 months) in metropolitan France, Central African Republic, and South America.
  Control subjects will be included in the hospital when they come for consultation for reasons other than diarrhea.
  Children suffering from acute or chronic diarrhea will be included in the hospital during a consultation.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Plasma levels of vitamin C | 1 year
  Plasma levels of vitamin C will be used to determine whether vitamin-deficiency may occurs in children living in developing countries

SECONDARY OUTCOMES:
Plasma levels of vitamin A, C and E | 1 year
  Plasma levels of vitamin A, C and E will be used to determine the plasma vitamin A, C and E concentrations in children suffering of diarrheal diseases

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Manirakiza, MD, PhD, Principal Investigator — Institut Pasteur de Bangui, Centrafrican Republic; Thomas Blanc, MD, PhD, Principal Investigator — Hopital Necker Paris, France; Jean-Chrysostome Gody, MD, PhD, Principal Investigator — Complexe Pédiatrique de Bangui, Centrafrican Republic; Emilie Huguon, MD, Principal Investigator — Centre Hospitalier Térritorial Gaston Bourret, New Caledonia
Locations (3):
- Complexe Pédiatrique, Bangui, Central African Republic
- Hopital Necker, Paris, France
- Centre Hospitalier Territorial Gaston Bourret, Noumea, New Caledonia

IPD SHARING:
Plan to Share IPD: No